CLINICAL TRIAL: NCT02917707
Title: Integrative Analysis of CRC Liver Metastasis
Acronym: CRC-LM
Status: Recruiting | Type: Observational
Sponsor: Da Fu (Other)
Collaborators: Ganzhou City People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Da Fu, Principal Investigator, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: Y219J11311
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Metastasis
Keywords: CRC; liver metastasis
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- normal colorectal tissues (PN): normal colorectal tissues
  Interventions: Other: normal colorectal tissues
- primary colorectal carcinoma tissues: primary colorectal carcinoma tissues
  Interventions: Other: normal colorectal tissues
- liver metastasis tissues: liver metastasis tissues
  Interventions: Other: normal colorectal tissues

INTERVENTIONS:
Other: normal colorectal tissues — The investigators will extract total protein, DNA and RNA from these groups.
  Other Names: primary colorectal carcinoma tissues; liver metastasis tissues

SUMMARY:
The investigators will perform integrative analysis of CRC liver metastasis

DETAILED DESCRIPTION:
The investigators will analyzed proteomes of paired normal colorectal tissues and colorectal cancer (CRC) with or without liver metastasis, sequenced transcriptomes, performed whole exome sequencing, and single nucleotide polymorphism (SNP) array profiling for triplets, each comprising normal colorectal tissue, primary colorectal carcinoma, and its synchronous matched liver metastasis, as well as analyzed genomics of CRC characterized previously by The Cancer Genome Atlas (TCGA) to conduct integrated proteogenomic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 75 years with histologically proven CRC
* No severe major organ dysfunction
* WHO performance status of 0 or 1
* No prior cancer chemotherapy

Exclusion Criteria:

* Age ≥ 76
* Severe major organ dysfunction
* World Health Organization (WHO) performance status of >1
* Prior cancer chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with CRC
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
5 years overall survival | 5 years

SECONDARY OUTCOMES:
5 years disease-free survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Da Fu, Ph.D., Principal Investigator — the Shanghai Tenth People's Hospital
Locations (2):
- China (2):
  - Ganzhou City People's Hospital, Ganzhou, Jiangxi
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
The investigators are willing to share data.

REFERENCES:
- [Result] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Derived] Ma YS, Huang T, Zhong XM, Zhang HW, Cong XL, Xu H, Lu GX, Yu F, Xue SB, Lv ZW, Fu D. Proteogenomic characterization and comprehensive integrative genomic analysis of human colorectal cancer liver metastasis. Mol Cancer. 2018 Sep 21;17(1):139. doi: 10.1186/s12943-018-0890-1. PMID 30241526